CLINICAL TRIAL: NCT04374890
Title: Evaluation of a New Supporting Ostomy Product
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CP308
Record Dates: First submitted 2020-04-29; First posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Stoma Ileostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Device: CP308

INTERVENTIONS:
Device: CP308 — 3 weeks of baseline followed by 2x3 weeks use of the test device

SUMMARY:
The aim of the study is to evaluate if the new supporting product influences wear time. It is the expectation that median wear time is slightly reduced in the period when subjects are using the supporting product with their ostomy appliance. Long-term benefits of the test product may be less skin redness, less worry of leakage and/or improvement in quality of life and social activities.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Be at least 18 years of age and have full legal capacity
3. Have had a stoma for more than three months
4. Have intact skin on the area used in the evaluation meaning no broken skin and only minor discoloration of the skin (assessed by investigator)
5. Be able to use one of the three test products (i.e. Ø50, Ø60 and Ø70 mm)
6. Have an ileostomy- or colostomy with liq-uid output (Bristol scale type 6-7)
7. Currently using a SenSura Mio product (1pc/2pc Flat/Convex/Concave)
8. Be willing and suitable (determined by the study nurse) to use the test product with-out using a paste/mouldable ring during the test periods
9. Have self-reported problems with leakage* (three times within 14 days) *Leakage: Leakage is defined as output from the stoma on the backside of the baseplate (underneath the baseplate)

Exclusion Criteria:

1. Currently receiving or have within the past 2 month received radio- and/or chemotherapy
2. Currently receiving or have within the past month received topical steroid treatment in the peristomal skin area or systemic steroid (tablet/injection) treatment
3. Are pregnant or breastfeeding
4. Participating in other interventional clinical investigations or have previously participat-ed in this investigation. Exception: Participation in other Coloplast sponsored clinical investigations is accepted under the circumstances that the subject has paused the activities in the investigation and are otherwise complying with the inclusion and exclusion criteria of this (CP308) protocol
5. Known sensitivity towards test product
6. Known sensitivity towards acrylate
7. Users with a pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Wear time | 9 weeks
  To evaluate the subject change pattern (wear time) when using the supporting product in 'real-life' situations'

CONTACTS AND LOCATIONS:
Locations (1):
- Coloplast A/S, Humlebæk, Denmark